CLINICAL TRIAL: NCT07209046
Title: A Randomized, Double-blind, Double-arm Study Conducted Directly With Consumers Via an App "Baritastic App", Evaluating the Efficacy of a Supplement Containing Bifidobacterium Lactis B420 and Pasteurized Akkermansia Muciniphila (UltraFlora® Triplebiotic) for 3 Months in Adults After Discontinuation of GLP-1 Treatment.
Brief Title: Impact of Probiotic (UltraFlora® Triplebiotic) on Weight Evolution on People After Discontinuation of GLP-1 Treatment.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Metagenics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GLO-NAM-2025-04
Record Dates: First submitted 2025-09-18; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Adults; GLP-1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UltraFlora® Triplebiotic (Active Comparator): The duration of trial intervention and participation for an individual participant is approximately 3 months (12 weeks). Screening, during which eligibility to participate in the trial is assessed, occurs at baseline. A fixed, orally administered, dose of the study products (UltraFlora® Triplebiotic, 2 capsules/day) are taken daily with breakfast.
  Interventions: Dietary Supplement: UltraFlora® Triplebiotic
- Orally administration of 2 capsules/day of placebo (Placebo Comparator): The duration of trial intervention and participation for an individual participant is approximately 3 months (12 weeks). Screening, during which eligibility to participate in the trial is assessed, occurs at baseline. A fixed, orally administered, dose of the placebo (2 capsules/day) are taken daily with breakfast.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: UltraFlora® Triplebiotic — The duration of trial intervention and participation for an individual participant is approximately 3 months (12 weeks). Screening, during which eligibility to participate in the trial is assessed, occurs at baseline. A fixed, orally administered, dose of probiotic ( UltraFlora® Triplebiotics, 2 capsules/day) are taken daily with a glass of water.
  Arms: UltraFlora® Triplebiotic
Dietary Supplement: Placebo — The duration of trial intervention and participation for an individual participant is approximately 3 months (12 weeks). Screening, during which eligibility to participate in the trial is assessed, occurs at baseline. A fixed, orally administered, dose of placebo (2 capsule/day) are taken daily with a glass of water.
  Arms: Orally administration of 2 capsules/day of placebo

SUMMARY:
This is a randomized, double-blind, double arm study involving 128 participants who will undergo a total participation period of 12 weeks.

DETAILED DESCRIPTION:
The trial begins with a screening to assess eligibility, followed by a 12-week treatment phase during which participants will receive a fixed-dose oral supplementation regimen. During this treatment period, participants will take UltraFlora® Triplebiotic at a fixed dose of 2 capsule per day, administered orally once daily with food. During the 12-week treatment period, participants will be asked to complete questions and track their weight changes.

ELIGIBILITY:
Inclusion Criteria:

1. Providing written informed consent
2. Males and females of at least 18 years old
3. Body mass index (BMI) between 25 and 30 (including 25 and 30) (Weight: 25 < BMI < 30)
4. Having undergone treatment with GLP-1 for more than 3 months but for less than 1 year.
5. Having stopped GLP-1 treatment for a maximum of 4 weeks
6. Being willing to maintain stable dietary habits and physical activity levels throughout the trial period
7. Being willing not to introduce any other food supplements during the trial period (supplements used in the two weeks prior to enrolling in the trial and used consistently throughout are acceptable, except for probiotics).

Exclusion Criteria:

1. Being on GLP-1 treatment
2. Having had any type of bariatric surgery, or planned bariatric surgery during the period of trial participation.
3. Suffering from a severe chronic disease (e.g., cancer, HIV, hepatic or renal impairment, diabetes type I), inflammatory bowel disease (IBD), Coeliac Disease, and/or being immunocompromised.
4. Suffering from any uncontrolled endocrine disorder.
5. Having consumed any probiotic supplements in the 3 months prior to enrollment.
6. Having used any antibiotic treatment in the 3 months prior to enrollment.
7. Having a known allergy to the ingredients in the study product.
8. Being pregnant or lactating (breastfeeding) or trying to become pregnant.
9. Participating in an other clinical trial.
10. Suffering from dementia or inability to take the trial treatment in an appropriate way.
11. Taking UltraFlora® Triplebiotic or any similar product from competitors prior to trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
weight measurement | From enrollment to the end of treatment at 12 weeks (90 days)
  Evaluate the impact of UltraFlora Triplebiotic (containing Bifidobacterium Lactis B420 and pasteurized Akkermansia Muciniphila) on weight regain over 3 months after discontinuation of GLP-1.

SECONDARY OUTCOMES:
IBS-SSS (Irritable Bowel Syndrome - Severity Scoring System) questionnaire | From enrollment to the end of treatment at 12 weeks (90 days)
  Evaluate the impact of UltraFlora Triplebiotic containing Bifidobacterium Lactis B420 and pasteurized Akkermansia Muciniphila on weight regain over 3 months after discontinuation of GLP-1. It is a visual analog scale ranging from 0 to 100 that allows the severity of patients' gastrointestinal symptoms to be assessed. The higher the score, the more pain the patient is experiencing.
SVS (Subjective Vitality Scale) questionnaire | From enrollment to the end of treatment at 12 weeks (90 days)
  Evaluate the impact of UltraFlora Triplebiotic containing Bifidobacterium Lactis B420 and pasteurized Akkermansia Muciniphila on vitality using the Subjective Vitality Scales (SVS) questionnaire. This questionnaire assesses a state of well-being and optimal functioning in relation to independence and physical and psychological health. Scores range from 1 (very low vitality) to 7 (optimal vitality).
TFEQ-R18 (Three-Factor Eating Questionnaire - Revised 18 items) Questionnaire | From enrollment to the end of treatment at 12 weeks (90 days)
  Evaluate the impact of UltraFlora Triplebiotic containing Bifidobacterium Lactis B420 and pasteurized Akkermansia Muciniphila on Hunger, Appetite and Cravings using the TFEQ-R18 Questionnaire over the course of 90 days. The TFEQ-R18 is a psychometric questionnaire that assesses eating behaviors and attitudes toward food. There are three dimensions: CR = conscious restraint, UE = uncontrolled eating, EE = emotional eating. High scores in UE or EE indicate an increased risk of overeating, weight gain, or eating disorders. A high score in CR shows a strong desire to restrict intake, but this is sometimes associated with episodes of disinhibition if the restriction fails.

OTHER OUTCOMES:
Assessment of appetite (e.g., number of meals) and food cravings (e.g., snacking or food preferences) in seven questions. | From enrollment to the end of treatment at 12 weeks (90 days)
  How hungry were you today? How full do you feel right now? How many meals ? Did you think about your next meal when you finished your meal? How many craving did you have today? How strong is your desire to eat? How much food do you think you could eat right now?
Side effects experienced when taking the test product or placebo throughout the study (product tolerance) | The proportion of participants at day 14 (T1), day 30 (T2), day 60 (T3), day 90 (T4),
  Expressed any of the following symptoms: headache(s), rash(es), cough, changes in appetite, or other.
patient satisfaction with product use and recommendation | The proportion of participants that at day 90 (T4):
  Evaluate the impact of UltraFlora Triplebiotic containing Bifidobacterium Lactis B420 and pasteurized Akkermansia Muciniphila after 90 days.
  Is satisfied with the intervention ? Would recommend the product ? Would purchase the product ?

CONTACTS AND LOCATIONS:
Overall Officials: Mieke Van Den Driessche, PhD, Study Director — Metagenics, Inc.; Irfan Qureshi, MD, Principal Investigator — Metagenics, Inc.

IPD SHARING:
Plan to Share IPD: No